CLINICAL TRIAL: NCT00898859
Title: Role of ADAMs in Epithelial Dysregulation in COPD. Differences Between From Non-smokers, Healthy Smokers and Patients With COPD.
Brief Title: Role of A Disintegrin and Metalloproteinase (ADAM) in Epithelial Dysfunction
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Maarten van den Berge, doctor, University Medical Center Groningen
Other Study IDs: METc2009086
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: ADAM; epithelial; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bronchial brushes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Healthy, non-smoking
- 2: healthy, ex-smoking
- 3: healthy, current-smokers
- 4: COPD, ex-smokers
- 5: COPD, smokers

SUMMARY:
Despite emerging implications for ADAMs (and matrix metalloproteinases (MMPs)) in disease progression, the mechanisms that lead to activation of specific ADAMs (and MMPs) and their actions in chronic obstructive pulmonary disease (COPD) are still incompletely understood. In the current study, the researchers aim to investigate the effects of cigarette smoke on cellular parameters that are relevant for development of COPD and the involvement of ADAM activity in these effects. By studying the effects of ADAM inhibition, the researchers aim to provide novel insights in the role of ADAMs in the development of COPD, which may offer new therapeutic targets for the treatment of COPD.

DETAILED DESCRIPTION:
Smoking is the largest risk factor for the development of COPD. It has been shown in patients with COPD that smoking induces airway inflammation characterized by bronchial infiltration of neutrophils, macrophages, lymphocytes and mast cells. In addition, smoking accelerates lung function loss and increases bronchial hyperresponsiveness, symptoms, and even mortality in COPD. When inhaled, tobacco smoke first encounters the airway epithelium, which forms a barrier to environmental substances and limits their access to the subepithelial layer. There is suggestive evidence that impaired repair responses and loss of epithelial integrity in the airways play a crucial role in the pathogenesis and contribute to tissue remodeling in COPD. Remodeling of the airway epithelium, e.g., squamous metaplasia and mucous hyperplasia, is often observed in COPD.

Metalloproteases (MMPs) and A Disintegrin and Metalloproteinase (ADAM)s may play an important role in respiratory diseases. MMPs and ADAMs, a class of membrane-bound MMPs, form a family of enzymes involved in degrading extracellular matrix (ECM) components. Their proteolytic activity is involved in remodeling of the ECM, which is required for migration and repair processes and regulated tissue turn-over. However, aberrant activity can lead to tissue destruction and irreversible damage. Thus MMPs, and ADAMs may play an important role in respiratory diseases and a protease-antiprotease imbalance may contribute to airway remodeling and impaired epithelial repair in COPD. In addition, MMPs/ADAMs act in regulatory events in inflammation and airway remodeling by liberating adhesion molecules and shedding of growth factors and cytokines from the cell surface. Furthermore, ADAMs play a role in cell-cell and cell-matrix interactions by their so-called disintegrin domain. In epithelial cells, both MMPs and ADAMs are known to regulate intercellular contacts, cell-matrix contacts, migratory responses, shedding of cytokines/growth factors, and intracellular signaling pathways. Since increased MMP levels (e.g., MMP-9, 12) have been observed during COPD exacerbations and polymorphisms in specific ADAM genes (i.e., ADAM33) have been associated with COPD susceptibility, the activation of MMPs and ADAMs on the airway epithelium may play an important role in the pathogenesis of COPD. Reactive oxygen species present in cigarette smoke may activate Duox, leading to activation of ADAM17 in airway epithelial cells. ADAM17 has been described to be involved in the release of growth factors (TGF-α), leading to the release of proinflammatory cytokines (IL-8) and production of MUC5AC 10-13. TGF-α acts on the EGF receptor (EGFR), which is involved in the production of MUC5AC and goblet cell hyperplasia. IL-8 is a well-known chemo-attractant for neutrophils, and thus may play a central role in neutrophilic inflammation in COPD, leading to ROS production, the release of neutrophil elastase and emphysema.

Despite emerging implications for ADAMs (and MMPs) in disease progression, the mechanisms that lead to activation of specific ADAMs (and MMPs) and their actions in COPD are still incompletely understood. In the current study, we aim to investigate the effects of cigarette smoke on cellular parameters that are relevant for development of COPD and the involvement of ADAM activity in these effects. By studying the effects of ADAM inhibition, we aim to provide novel insights in the role of ADAMs in the development of COPD, which may offer new therapeutic targets for the treatment of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years.
* Individuals who currently smoke ≥ 10 cigarettes/day and > 10 pack years.
* Documented FEV1 > 80% predicted, FEV1/FVC > 70%.
* Referred by own physician for a bronchoscopy.

Exclusion Criteria:

* Any disease that, as judged by the Investigator, could affect the outcome of this study.
* A respiratory tract infection within 4 weeks of the start of the study.
* History of myocardial infarction or documented myocardial ischemia or the presence of an artificial heart valve.
* Use of anticoagulants.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and subjects with COPD
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
IL8-production | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berge, PhD, Study Chair — University Medical Center Groningen; maarrten van den Berge, PhD, Study Director — University Medical Center Groningen; Irene Heijink, PhD, Principal Investigator — University Medical Center Groningen